CLINICAL TRIAL: NCT03593226
Title: A Phase I/IIa, Multicentre, Two Parts, Open-Label Study Designed to Evaluate the Safety and Tolerability of Escalating Doses of AGI-134 in Unresectable/Metastatic Solid Tumours
Brief Title: Study to Evaluate Safety & Tolerability of AGI-134 in Solid Tumour
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Agalimmune Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGI-134.FIM.101
Record Dates: First submitted 2018-06-05; First posted 2018-07-20 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Superficial, Palpable, Unresectable/Metastatic Solid Tumour

STUDY DESIGN:
Intervention Model Description: Part 1 (Accelerated escalation): An accelerated escalation dose study designed to assess the safety and tolerability of escalating doses of AGI-134, as well as the Maximum Tolerated Dose (MTD) and the Part 2 dose (RP2D).
  Part 2: This part of the study was designed to assess the safety, tolerability and anti-tumour activity of AGI-134 as a monotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AGI-134 25 mg (Experimental): 25 mg AGI-134 (1 mL) via intratumor injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
  Interventions: Drug: AGI-134
- AGI-134 50 mg (Experimental): 50 mg AGI-134 (2 mL) via intratumor injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
  Interventions: Drug: AGI-134
- AGI-134 100 mg (Experimental): 100 mg AGI-134 (4 mL) via intratumor injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
  Interventions: Drug: AGI-134
- AGI-134 200 mg (Experimental): 200 mg AGI-134 (8 mL) via intratumor injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
  Interventions: Drug: AGI-134

INTERVENTIONS:
Drug: AGI-134 — AGI-134 via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.

SUMMARY:
This study will evaluate if AGI-134 given alone is safe and tolerate in treating patients with unresectable/metastatic solid tumours.

DETAILED DESCRIPTION:
Study AGI-134.FIM.101 was a Phase I/IIa, first in man (FIM), multi-center, single-arm, open-label study, designed to evaluate the safety and tolerability of escalating doses of AGI-134 as a monotherapy in unresectable/metastatic solid tumors.

The study comprised of 2 parts:

Part 1 was an accelerated escalation of the AGI-134 dose, designed to assess the safety and tolerability of AGI-134, as well as to determine the MTD (maximum tolerated dose) and recommended dose for Part 2 of the study (RP2D).

Part 2 was designed to assess the safety, tolerability and biological activity of AGI-134 at the RP2D in subjects with either deep or superficial unresectable/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria

1. Adult male or female aged 18 years old or older.
2. Have a histologically or cytologically confirmed unresectable metastatic solid tumour and who have received or been intolerant to all curative treatment options and treatments demonstrated to prolong survival.
3. Subjects should have at least two measurable lesions based on RECIST v1.1 as determined by the site study team.
4. Subjects who are willing to undergo tumour biopsies, unless tumour is considered inaccessible or biopsy is otherwise considered not in the subject's best interest.
5. With sufficient tumour size for IT injection
6. Has ≥ 2 lesions:

   Has ≥1 injectable lesion which is amenable to injection and biopsy and is measurable according to RECIST v1.1.

   Has ≥1 metastatic lesion is amenable for biopsy and measurable according to RECIST v1.1
7. Evaluable Disease according to RECIST v1.1
8. Has an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
9. Has a life expectancy >3 months
10. Adequate organ function
11. Women of childbearing potential and all men must agree to use 2 methods of an adequate contraception
12. Subject is able and willing to comply with the requirements of the protocol.
13. Subject is able to voluntarily provide written informed consent.

Exclusion Criteria:

1. Has a disease that is suitable for therapy administered with curative intent.
2. Has any active, acute, or chronic infection(s) that are uncontrolled and/or requiring treatment, such as antibiotics
3. An active autoimmune disease that has required systemic treatment in the 2 years preceding the study
4. History of or plan for splenectomy or splenic irradiation
5. History of organ transplant or currently taking active immunosuppressive therapy
6. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
7. Has known active or chronic Hepatitis B or Hepatitis C
8. History or evidence of cancer associated with immunodeficiency states
9. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
10. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
11. Is expected to require any other form of antineoplastic therapy while on study
12. Had received live vaccines within 30 days prior to the first dose of trial treatment.
13. Has positive Immunoglobulin E (IgE) anti -Gal
14. Subject has a known allergy to alpha-Gal, such as red meat allergy, exposure to lone star tick (Amblyomma americanum), Ixodes ricinus/ holocyclus, or Cetuximab allergy
15. Has known allergy or hypersensitivity to any of the test compounds, materials or contraindication to test product
16. History or evidence of central nervous system metastases and/or carcinomatous meningitis (unless stable without treatment for at least 6 weeks and not requiring steroids)
17. Has received other experimental therapies or used an investigational device within 28 days of the first dose of treatment
18. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 14 days prior to study Day 1 or has not recovered from Adverse Event (AE) ≤ Grade 1 by treatment administered more than 14 days before first dose
19. Has had a prior anti-cancer monoclonal antibody (mAb) within 28 days prior to study Day 1 or who has not recovered from AE ≤ Grade 1 by treatment administered more than 28 days earlier.
20. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
21. Has unstable angina, new onset angina within the last 3 months, myocardial infarction within the last 6 months, uncontrolled atrial fibrillation, or current congestive heart failure with New York Heart Association Class III or higher.
22. Has a known current additional malignancy that is progressing or requires active treatment
23. O2 saturation < 92% (on room air).
24. Has an underlying medical condition that would preclude study participation or other psychological, social or physical examination finding or a laboratory abnormality that the Investigator considers would make the subject a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
25. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (3):
  - UCLA, Los Angeles, California
  - AHS Hospital Corp., Morristown, New Jersey
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
- Israel (5):
  - Emek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- United Kingdom (6):
  - University of Birmingham, Birmingham
  - Edinburgh Cancer Research Centre, Edinburgh
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - University Collage London, London
  - The Christie NHS Foundation Trust, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AGI-134 25 mg: 25 mg AGI-134 (1 mL) via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
- AGI-134 50 mg: 50 mg AGI-134 (2 mL) via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
- AGI-134 100 mg: 100 mg AGI-134 (4 mL) via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
- AGI-134 200 mg: 200 mg AGI-134 (8 mL) via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
Period: Overall Study
Arm/Group | AGI-134 25 mg | AGI-134 50 mg | AGI-134 100 mg | AGI-134 200 mg
Started | 6 | 19 | 7 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 19 | 7 | 6
Not completed — Disease progression | 6 | 13 | 5 | 6
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 4 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Clinical disease progression | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set - all enrolled subjects in each specific dose
Groups:
- AGI-134 25mg/1mL: AGI-134 1mL via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
- AGI-134 50mg/2mL: AGI-134 2mL via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
- AGI-134 100mg/4mL: AGI-134 4mL via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
- AGI-134 200mg/8mL: AGI-134 8mL via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists in three weeks, dosing will be given for 4 cycles.
- Total: Total of all reporting groups
Arm/Group | AGI-134 25mg/1mL | AGI-134 50mg/2mL | AGI-134 100mg/4mL | AGI-134 200mg/8mL | Total
Number analyzed (Participants) | 6 | 19 | 7 | 6 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 11 | 5 | 3 | 20
  >=65 years | 5 | 8 | 2 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (8.2) | 59.95 (13.4) | 54 (11) | 59.2 (18.5) | 60 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 2 | 3 | 17
  Male | 5 | 8 | 5 | 3 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 6 | 19 | 6 | 5 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 12 | 6 | 4 | 24
  Israel | 2 | 3 | 0 | 0 | 5
  Spain | 2 | 4 | 1 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of AGI-134 Injected Intra-tumourally (IT)
Description: Safety and tolerability of AGI-134 injected intra-tumourally (IT) by assessment of the percentage of participants who experienced a dose-limiting toxicity (DLT) . DLTs will be assessed during the first cycle (21 days)
Time Frame: Up to 3 weeks after first administration of each dose level
Measure: Count of Participants; unit: Participants
Groups:
- AGI-134 25 mg: 25 mg AGI-134 (1 mL) via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists of three weeks, dosing will be given for 4 cycles.
- AGI-134 50 mg: 50 mg AGI-134 (2 mL) via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists of three weeks, dosing will be given for 4 cycles.
- AGI-134 100 mg: 100 mg AGI-134 (4 mL) via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists of three weeks, dosing will be given for 4 cycles.
- AGI-134 200 mg: 200 mg AGI-134 (8 mL) via IT injection. The proposed treatment is one dose of AGI-134 monotherapy per cycle; each cycle consists of three weeks, dosing will be given for 4 cycles.
Arm/Group | AGI-134 25 mg | AGI-134 50 mg | AGI-134 100 mg | AGI-134 200 mg
Number analyzed (Participants) | 6 | 19 | 7 | 6
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Discontinue Study Drug Due to an Adverse Events
Description: Percentage of Participants Who Discontinue Study Drug Due to an Adverse Event (AE) AEs are defined as any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of the study treatment, is also an AE. The percentage of participants who discontinue study treatment due to an AE will be presented
Time Frame: Approximately 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | AGI-134 25mg/1mL | AGI-134 50mg/2mL | AGI-134 100mg/4mL | AGI-134 200mg/8mL
Number analyzed (Participants) | 6 | 19 | 7 | 6
Participants | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs collected during the course of the study from Informed Consent Form (ICF) signature time until study completed or ceased, approximately 12 months.
Groups:
- Overall: Safety Population (all treated participants)
Arm/Group | Overall | AGI-134 25 mg | AGI-134 50 mg | AGI-134 100 mg | AGI-134 200 mg
All-Cause Mortality (participants affected / at risk) | 1/38 | 0/6 | 0/19 | 0/7 | 1/6
Serious Adverse Events (participants affected / at risk) | 18/38 | 3/6 | 8/19 | 2/7 | 5/6
Other Adverse Events (participants affected / at risk) | 38/38 | 6/6 | 19/19 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=38) | AGI-134 25 mg (N=6) | AGI-134 50 mg (N=19) | AGI-134 100 mg (N=7) | AGI-134 200 mg (N=6)
Catheter site infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall (N=38) | AGI-134 25 mg (N=6) | AGI-134 50 mg (N=19) | AGI-134 100 mg (N=7) | AGI-134 200 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 7 (15) | 1 (1) | 4 (12) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (8) | 0 (0) | 3 (3) | 0 (0) | 2 (5)
Dyspepsia (Gastrointestinal disorders) | 3 (5) | 1 (1) | 1 (3) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (5) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (6) | 0 (0) | 2 (3) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 9 (14) | 1 (3) | 4 (5) | 2 (2) | 2 (4)
Vomiting (Gastrointestinal disorders) | 11 (16) | 0 (0) | 6 (8) | 2 (3) | 3 (5)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parotid gland haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tongue movement disturbance (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 14 (22) | 3 (3) | 6 (13) | 4 (5) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 5 (10) | 0 (0) | 3 (4) | 0 (0) | 2 (6)
Chills (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site discharge (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site discomfort (General disorders) | 2 (4) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Injection site oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 10 (13) | 2 (3) | 2 (2) | 3 (4) | 3 (4)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nodule (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (5) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Activated partial thromboplastin time shortened (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Past-pointing (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood albumin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 4 (6) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Protein urine present (Investigations) | 2 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (9) | 0 (0) | 6 (6) | 1 (2) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (10) | 1 (1) | 3 (5) | 1 (2) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (1) | 1 (5) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 0 (0) | 1 (5) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (8) | 0 (0) | 2 (4) | 1 (3) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 8 (9) | 1 (1) | 5 (6) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Libido increased (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder dilatation (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract discomfort (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (11) | 1 (1) | 4 (6) | 3 (4) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 3 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Systolic hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The restrictions are as per the signed agreement with each PI and institution.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT03593226/Prot_SAP_000.pdf